CLINICAL TRIAL: NCT07096323
Title: Successful Treatment of Female Pattern Hair Loss With Non-Cultured Adipose Derived Stem Cells (ADSCs) in Mechanically Emulsified Adipose Tissue (Nanofat) With and Without Platelet-Rich Plasma (PRP): A Randomized Clinical Trial
Brief Title: Successful Treatment of Female Pattern Hair Loss With Injection of Nanofat With and Without Platelet-Rich Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS 167/2023; Does not exist (Other: Does not exist)
Record Dates: First submitted 2025-06-29; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-02

CONDITIONS: Female Pattern Hair Loss
Keywords: Adipose Derived Stem Cells; Nanofat; Platelet Rich Plasma

STUDY DESIGN:
Intervention Model Description: The study included 40 patients with FPHL. Patients were divided into two groups (20 patients each) using simple (computer-generated) randomization. Group A: Nanofat was prepared and injected intradermally into the frontoparietal scalp. Group B: Nanofat was prepared, then mixed with PRP, and injected as in group A.
  A single session was performed for patients in both groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nanofat only (Active Comparator): 20 patients received a single session of scalp injection with nanofat only.
  Interventions: Procedure: Nanofat only
- Nanofat mixed with PRP (Active Comparator): 20 patients received a single session of scalp injection with nanofat mixed with PRP.
  Interventions: Procedure: Nanofat mixed with PRP

INTERVENTIONS:
Procedure: Nanofat only — Fat was collected from either the lower abdomen or lateral upper thigh. A blunt-tipped infiltration cannula (Luer Lock Mercedes Gold Liposuction Cannula 4mm x 30 cm, Pakistan) was used for injection of Klein solution for tumescent anesthesia. Liposuction cannula was then used, connected to a 50 ml syringe mounted with a stopper to generate negative pressure for liposuction. The lipoaspirate was washed to obtain pure adipose tissue, and mechanical emulsification was achieved by transferring the fat through progressively smaller sieves (2.2 mm, 1.5 mm, 1.2 mm) between two 10 ml syringes connected with Luer-Lock connectors, with at least 30 passages each. The emulsion was not filtered and is referred to as "Nanofat 2.0."
  Arms: Nanofat only
Procedure: Nanofat mixed with PRP — Nanofat is prepared the same way as arm 1. PRP was prepared as follows: Ten milliliters of venous autologous whole blood were collected with tri-sodium citrate as an anticoagulant, then centrifuged at 112g (1000 rpm) for 10 minutes. The plasma was transferred to new tubes without tri-sodium citrate and centrifuged again at 448g (2000 rpm) for 10 minutes to separate the platelet pellet and platelet-poor plasma (PPP). PRP was kept for mixing it with nanofat while PPP was discarded
  Arms: Nanofat mixed with PRP

SUMMARY:
Background: FPHL is a chronic progressive condition that necessitates lifelong management. Over time, patients who respond to conventional therapy may experience a decrease in the effectiveness of their treatment and may require alternative interventions to delay disease progression and enhance the efficacy of current therapies. ADSCs have demonstrated potential as a regenerative interventional modality for the treatment of such conditions.

Objective: To compare efficacy of nanofat alone and nanofat combined with platelet-rich plasma (PRP) for the treatment of female-pattern hair loss.

Methods: This study is a randomized controlled prospective intervention. Forty patients with mild to moderate FPHL were selected and randomly allocated into two groups (A and B). Both groups received a single session of nanofat scalp injection. Nanofat was prepared from lipoaspirates by mechanical agitation of adipose tissue, and was mixed with PRP for patients allocated in group B.

Results: Nanofat alone and combined with PRP promoted hair regrowth. However, the adjunctive use of PRP with nanofat yielded a statistically significant enhancement in terminal hair thickness (P <0.001) and count (P <0.001) compared with nanofat alone. Mean satisfaction score was 3 out of 5 at 24 weeks post-injection, with no significant difference between the two treatment groups (P= 0.937). The side effects were mild and well-tolerated.

Conclusion: Both nanofat, alone and in combination with PRP, improved hair thickness and count in patients with FPHL. The combination with PRP demonstrated a statistically significant improvement compared with nanofat alone.

DETAILED DESCRIPTION:
Patients and Methods This randomized controlled clinical trial was conducted on 40 female patients presenting with pattern hair loss, selected from the outpatient clinic of Dermatology, Venereology, and Andrology Department, Ain Shams University Hospitals, between December 2022 and July 2023.

Following approval from the research ethics committee of the Faculty of Medicine, Ain Shams University (FMASU MS 167/2023), written informed consent was obtained from each patient after providing information regarding procedural steps and potential side effects or complications.

The study population comprised females aged 18-50 years with moderate to severe FPHL, classified as Sinclair grades 3-4. Exclusion criteria included age < 18 years and >50 years, chronic telogen effluvium, use of topical or systemic FPHL treatments in the preceding 6 months, infection at the treatment site or elsewhere, diabetes, hemorrhagic disorders, anticoagulant therapy, pregnancy or lactation, personal or family history of malignancy, immunosuppression or lidocaine allergy.

The clinical diagnosis of FPHL was confirmed according to Rakowska et al., 2009 trichoscopic criteria for diagnosis of FPHL. FPHL is diagnosed by the presence of two major criteria or one major and two minor criteria.

Digital photography was documented at a point 10 cm directly above the midpoint of the glabella at the initial visit and at all subsequent visits. Patients were evaluated clinically and trichoscopically at baseline, then at 12 and 24 weeks after treatment.

Patients were divided into two groups (20 patients each) using simple (computer-generated) randomization. Group A: Nanofat was prepared and injected intradermally into the frontoparietal scalp. Group B: Nanofat was prepared, then mixed with PRP, and injected as in group A.

A single session was performed for patients in both groups. Nanofat Preparation: Fat was collected from either the lower abdomen or lateral upper thigh. A blunt-tipped infiltration cannula (Luer Lock Mercedes Gold Liposuction Cannula 4mm x 30 cm, Pakistan) was used for injection of Klein solution for tumescent anesthesia. Liposuction cannula was then used, connected to a 50 ml syringe mounted with a stopper to generate negative pressure for liposuction. The lipoaspirate was washed to obtain pure adipose tissue, and mechanical emulsification was achieved by transferring the fat through progressively smaller sieves (2.2 mm, 1.5 mm, 1.2 mm) between two 10 ml syringes connected with Luer-Lock connectors, with at least 30 passages each. The emulsion was not filtered and is referred to as "Nanofat 2.0." PRP preparation: Ten milliliters of venous autologous whole blood were collected with tri-sodium citrate as an anticoagulant, then centrifuged at 112g (1000 rpm) for 10 minutes. The plasma was transferred to new tubes without tri-sodium citrate and centrifuged again at 448g (2000 rpm) for 10 minutes to separate the platelet pellet and platelet-poor plasma (PPP). PRP was kept for mixing it with nanofat while PPP was discarded.

Evaluation of the results The results were evaluated using the following assessments. A- Clinical Evaluation: Clinical photographs of the centrally parted scalp were taken with an iPhone 13 Pro Max camera 12-megapixel camera, ensuring standardization in light, angle, and position. Two blinded investigators evaluated hair fullness and clinical grade using the Sinclair classification and Investigator Global Assessment (IGA) scale, ranging from -1 (worsening) to 3 (excellent improvement).

B- Trichoscopic Examination: Trichoscopic images were obtained using a Dermlite DLIII dermoscope (3Gen Inc., California, USA) at 10x magnification. They were analysed using a simple morphometric software (ImageJ, National Institutes of Health, Bethesda, Maryland, USA) to manually count and measure the mean diameter of terminal hairs.

C- Patient Satisfaction: Patients completed a 5-point Likert scale questionnaire to assess their subjective satisfaction with changes in hair density, hair quality and hair fall at week 24.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-50 years with moderate to severe FPHL, classified as Sinclair grades 2-4.

Exclusion Criteria:

* Age less than 18 years or more than 50 years
* Chronic telogen effluvium
* Use of topical or systemic FPHL treatments in the preceding 6 months
* Infection at the treatment site or elsewhere
* Uncontrolled iabetes, hemorrhagic disorders, anticoagulant therapy, pregnancy or lactation
* Personal or family history of malignancy, immunosuppression or lidocaine allergy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female pattern hair loss is a condition that affects females only.
Enrollment: 40 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Increase in terminal hair count | 24 weeks
  After treatment with ADSCs, the anticipated primary outcome measure is trichoscopic increase in terminal hair count. This was compared with nanofat alone versus mixed with PRP.
Increase in terminal hair thickness | 24 weeks
  After treatment with ADSCs, the anticipated primary outcome measure is trichoscopic increase in terminal hair thickness. This was compared with nanofat alone versus mixed with PRP.

CONTACTS AND LOCATIONS:
Overall Officials: Mahy El-Bassiouny, Study Director — Ain Shams University
Locations (1):
- Dermatology Department- Ain Shams University, Cairo, Egypt